CLINICAL TRIAL: NCT04846309
Title: Hypoxia Imaging for Esophageal Cancer to Guide Personalized Radiation Therapy
Acronym: PIONEER
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University of Utah (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HCI137650
Record Dates: First submitted 2021-04-12; First posted 2021-04-15 (Actual); Last update posted 2025-05-07 (Actual); Status verified 2025-05

CONDITIONS: Esophageal Cancer
MeSH Terms: conditions — Esophageal Neoplasms | interventions — Radiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment: all patients (Experimental)
  Interventions: Radiation: Radiation; Drug: FMISO PET CT

INTERVENTIONS:
Radiation: Radiation — Prior to the start of study therapy, eligible subjects will receive a FMISO-PET scan. If there is uptake visualized on the scan, the tumor will be considered as hypoxic. If there is no uptake seen on the FMISO-PET scan, tumors will be labeled not hypoxic. Subjects with tumors identified by imaging as hypoxic will be treated with a higher dose of radiation therapy. Tumors will be defined as being hypoxic if FMISO accumulation occurs as demonstrated by standardized uptake value (SUV) uptake in the tumor.
Drug: FMISO PET CT — Prior to the start of study therapy, eligible subjects will receive a FMISO-PET scan. If there is uptake visualized on the scan, the tumor will be considered as hypoxic. If there is no uptake seen on the FMISO-PET scan, tumors will be labeled not hypoxic.

SUMMARY:
This is a Phase I trial evaluating the safety of personalized radiation therapy based on levels of hypoxia identified on FMISO-PET and MRI. All patients will receive a baseline FMISO positron emission tomography (PET) and MRI to identify levels of hypoxia. Patients with tumor hypoxia will receive a higher dose of radiation therapy. Subjects who do not have hypoxic tumors will be treated with the standard-of-care radiation regimen. After fraction 10 of radiation therapy, an additional MRI will be performed. If this interim MRI demonstrates little or no response (as defined in Section 6), an optional boost radiation dose can be administered.

Trial enrollment will be conducted in two parts. In Part 1, eight patients will be enrolled. After all eight patients have completed the 30 day dose-limiting toxicity (DLT) period, enrollment will be placed on hold and safety will be evaluated. During the interim analysis, one additional patient will be allowed to be enrolled in the trial. If the trial meets stopping rules as described in Section 11.3, the trial will be re-evaluated by the Data and Safety Monitoring Committee (DSMC) and the Principal Investigator. However, if the rate of DLTs remains below the unacceptable toxicity rate, enrollment will open to the enrollment of eight more patients.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subject aged ≥ 18 years.
* Esophageal cancer patient eligible to undergo either neoadjuvant or definitive chemoradiation therapy (CRT).

Note: Stage IV patients with limited metastatic disease burden may be eligible if CRT is recommended by the multidisciplinary team.

* Eastern Cooperative Oncology Group (ECOG) Performance Status ≤ 2.
* For female subjects: Negative pregnancy test or evidence of post-menopausal status. The post-menopausal status will be defined as having been amenorrheic for 12 months without an alternative medical cause. The following age-specific requirements apply:

  * Women < 50 years of age:

    * Amenorrheic for ≥ 12 months following cessation of exogenous hormonal treatments; and
    * Luteinizing hormone and follicle-stimulating hormone levels in the post-menopausal range for the institution; or
    * Underwent surgical sterilization (bilateral oophorectomy or hysterectomy).
  * Women ≥ 50 years of age:

    * Amenorrheic for 12 months or more following cessation of all exogenous hormonal treatments; or
    * Had radiation-induced menopause with last menses >1 year ago; or
    * Had chemotherapy-induced menopause with last menses >1 year ago; or
    * Underwent surgical sterilization (bilateral oophorectomy, bilateral salpingectomy, or hysterectomy).
* Recovery to baseline or ≤ Grade 2 CTCAE v5 from toxicities related to any prior treatments, unless AE(s) are clinically non-significant and/or stable on supportive therapy.
* Able to provide informed consent and willing to sign an approved consent form that conforms to federal and institutional guidelines.

Exclusion Criteria:

* Unable to undergo an MRI for any reason, including:

  * Severe claustrophobia not amenable to pre-medication
  * Presence of metallic objects or implanted medical devices in the body that are not MRI-compatible (e.g., non-MRI-compatible cardiac pacemaker, deep brain stimulator, neurostimulator, aneurysm clips, surgical clips, prostheses, artificial hearts, valves with steel parts, metal fragments, shrapnel, tattoos near the eye, or steel implants)
* Patients with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the radiation therapy are eligible for this trial.
* The subject has severe, uncontrolled, significant intercurrent or recent illness that would exclude them from being a candidate for chemoradiation therapy.

  --Any other condition that would, in the Investigator's judgment, contraindicate the subject's participation in the clinical study due to safety concerns or compliance with clinical study procedures.
* Known HIV infection with a detectable viral load at the time of screening. Note: Patients on effective antiretroviral therapy or who will plan on going on antiretroviral therapy at the time of screening are eligible for this trial. HIV testing is not required for eligibility.
* Known prior severe hypersensitivity to gadolinium, FMISO or any component in its formulations (NCI CTCAE v5.0 Grade ≥ 3).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2021-10-12 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
rate of grade ≥ 4 esophageal adverse events attributed to radiation therapy that occur within 30 days of finishing radiation therapy | 30 days after last study therapy
  assess the safety and tolerability of using hypoxia PET/CT imaging with Fluorine-18 fluoromisonidazole (FMISO) and MRI measures of radioresistance to personalize radiation therapy by delivering a higher dose of radiation to hypoxic tumors
rate of grade ≥ 4 esophageal adverse events attributed to radiation therapy that occur within 84 days of finishing radiation therapy | 84 days after last study therapy
  assess the safety and tolerability of using hypoxia PET/CT imaging with Fluorine-18 fluoromisonidazole (FMISO) and MRI measures of radioresistance to personalize radiation therapy by delivering a higher dose of radiation to hypoxic tumors
frequency of adverse events (AEs) and serious adverse events (SAEs) characterized by type, severity (as defined by the NIH CTCAE, version 5.0), seriousness, duration, and relationship to study treatment | 84 days after last study therapy
  assess the safety and tolerability of using hypoxia PET/CT imaging with Fluorine-18 fluoromisonidazole (FMISO) and MRI measures of radioresistance to personalize radiation therapy by delivering a higher dose of radiation to hypoxic tumors

SECONDARY OUTCOMES:
Progression-free survival (PFS) | Time from study therapy initiation to the time documented disease progression (as assessed by RECIST 1.1) or death from any cause for up to 18 months after last dose of study therapy
  assess the efficacy of hypoxia imaging-guided radiation treatment
Pathological complete response (pCR) rate | Long term follow up to occur for up to 18 months after last dose of study therapy.
  assess the efficacy of hypoxia imaging-guided radiation treatment

CONTACTS AND LOCATIONS:
Overall Officials: Shane Lloyd, MD, Principal Investigator — Huntsman Cancer Institute
Locations (1):
- Huntsman Cancer Institute, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No